CLINICAL TRIAL: NCT02053766
Title: Anesthesia in Patients With Mitochondrial Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to covid-19 we were not on track with enrollment rate
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maria Matuszczak, ◦Professor of Anesthesiology-Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HSC-MS-13-0600
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Results first posted 2024-07-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Mitochondrial Diseases
Keywords: Mitochondrial Diseases; Sevoflurane; Dexmedetomidine (Precedex®); Propofol
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Sevoflurane; Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane (Active Comparator): In the Operating Room (OR) after applying routine monitors, anesthesia will be induced with a mask using Sevoflurane up to 8%. Sevoflurane will be used for maintenance for the rest of the procedure with dosage between 1.5% and 4%. Vitals will be monitored. Fentanyl will be used as needed. Rocuronium will be used as needed for muscle relaxation. At the end of the procedure twitches will be evaluated and muscle relaxation will be reversed. Sevoflurane will be turned off at the end of procedure.
  Interventions: Drug: Sevoflurane
- Dexmedetomidine (Precedex®) (Active Comparator): These subjects will receive Dexmedetomidine intravenously. In the OR routine monitors will be placed. Vitals will be monitored. A loading dose of Precedex 1mcg/ kg will be given over 10 minutes. Infusion will be started using Precedex 1mcg/ kg/ hr and can be increased or decreased as needed. Fentanyl will be used as needed. Rocuronium will be used as needed for muscle relaxation. At the end of the procedure twitches will be evaluated and muscle relaxation will be reversed. Precedex infusion will be stopped at the end of the procedure.
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): These subjects will receive propofol for anesthesia maintenance. In the OR routine monitors will be placed. Vitals will be monitored. A loading dose of Propofol 2mg/ kg will be given over 2 minutes. Infusion will be started using Propofol 50 mcg/ kg/min and can be increased or decreased as needed (range 50-300mcg/kg/min). Fentanyl will be used as needed. Rocuronium will be used as needed for muscle relaxation. At the end of the procedure twitches will be evaluated and muscle relaxation will be reversed. Propofol infusion will be stopped at the end of the procedure.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane up to 8% will be administered to study subjects
  Other Names: Ultane
  Arms: Sevoflurane
Drug: Dexmedetomidine — Dexmedetomidine (Precedex) infusion starting at 1mcg/ kg/ hr will be administered to study subjects.
  Other Names: Precedex
  Arms: Dexmedetomidine (Precedex®)
Drug: Propofol — Propofol up to 50 mcg/ kg/min will be administered to study subjects.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
This pilot study is a prospective, randomized clinical trial to evaluate the effect of anesthesia in the mitochondrial dysfunction patient.

DETAILED DESCRIPTION:
Study subjects undergoing a routine medical care non-emergent procedure will be randomized into three different groups to receive one of the following anesthetic agents; Sevoflurane, Propofol or Dexmedetomidine.

The primary outcome of this pilot study is to evaluate and compare the incidence of adverse events in mitochondrial patients undergoing a diagnostic or therapeutic procedure up to 48 hours post anesthesia. The secondary outcome is to compare the metabolic derangements between three study groups by comparing changes in blood sugar, serum pH, serum bicarbonate, serum lactate and serum pyruvate levels before, during and after anesthesia in the groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfill the following inclusion criteria:
* Subject is informed and given ample opportunity to consider his/her participation and has given his/her written consent.
* Subject is willing and able to comply with all study requirements.
* Subject is between 0 - 17 years of age.
* Subject has been diagnosed with mitochondrial dysfunction based on modified Walker criteria.
* Subject is scheduled to have a non-emergent diagnostic or therapeutic procedure for routine medical care requiring general anesthesia estimated to last at least one hour.
* Subject is classified ASA I - IV

Exclusion Criteria:

Subjects are not permitted to enroll in the study if any of the following criteria are met:

* Subject is older than 17 years
* Subject is pregnant
* Subject is a nursing female and
* Subject has participated in the same study within 48 hours
* Subject is allergic or has had any adverse effect to any of the study agents in the past
* Anesthesia time is less than one hour
* Subject is classified ASA V

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Matuszczak, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sevoflurane | Dexmedetomidine (Precedex®) | Propofol
Started | 6 | 7 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Dexmedetomidine (Precedex®) | Propofol | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.5 (4.22) | 6.57 (4.15) | 4.33 (2.33) | 5.84 (3.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 5 | 5 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Time Frame: Up to 48 hours post anesthesia.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 7 | 6 | 6
Participants | 2 | 2 | 3

2. Secondary Outcome: Blood Glucose Level
Time Frame: Baseline
Population: Data were not collected for one participant in the Dexmedetomidine (Precedex®) arm. Data were not collected for one participant in the Propofol arm.
Measure: Mean (Standard Deviation); unit: milligrams per decilitre
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 6 | 5 | 6
milligrams per decilitre | 88.66 (15.29) | 89.20 (4.76) | 83.66 (10.2)

3. Secondary Outcome: Blood Glucose Level
Time Frame: 24 hours post-operative
Population: Data were not collected for 4 participants in the Dexmedetomidine (Precedex®) arm. Data were not collected for 4 participants in the Propofol arm. Data were not collected for 2 participants in the Sevoflurane arm.
Measure: Mean (Standard Deviation); unit: milligrams per decilitre
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 3 | 2 | 4
milligrams per decilitre | 87 (7) | 81.50 (13.43) | 93.75 (16.50)

4. Secondary Outcome: Serum pH
Description: The pH scale measures how acidic of alkaline a substance is and ranges from 0 to 14, where 7 is neutral, 14 is the most alkaline and 0 is the most acidic.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 6 | 5 | 6
score on a scale | 7.39 (7.37) | 7.36 (0.05) | 7.37 (0.02)

5. Secondary Outcome: Serum pH
Description: as for outcome 4
Time Frame: 24 hours post-operative
Population: Data were not collected for 4 participants in the Dexmedetomidine (Precedex®) arm. Data were not collected for 5 participants in the Propofol arm. Data were not collected for 4 participants in the Sevoflurane arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 3 | 1 | 2
score on a scale | 7.36 (0.05) | 7.40 (NA) — Standard Deviation not available since only 1 participant was analyzed for the assessment | 7.32 (0.04)

6. Secondary Outcome: Serum Bicarbonate
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 6 | 5 | 6
millimoles per liter | 25.50 (1.91) | 24.04 (3.66) | 25.23 (2.51)

7. Secondary Outcome: Serum Bicarbonate
Time Frame: 24 hours post-operative
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 3 | 1 | 2
millimoles per liter | 24.33 (4.16) | 20 (NA) — Standard Deviation not available since only 1 participant was analyzed for the assessment | 26.5 (2.12)

8. Secondary Outcome: Serum Lactate
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 6 | 5 | 6
millimoles per liter | 1.28 (0.44) | 0.82 (0.25) | 1.36 (0.58)

9. Secondary Outcome: Serum Lactate
Time Frame: 24 hours post-operative
Population: Data were not collected for 3 participants in the Dexmedetomidine (Precedex®) arm. Data were not collected for 3 participants in the Propofol arm. Data were not collected for 2 participants in the Sevoflurane arm.
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 4 | 3 | 4
millimoles per liter | 2.76 (0.47) | 1.15 (0.36) | 2.50 (0.65)

10. Secondary Outcome: Serum Pyruvate
Time Frame: Baseline
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligrams per decilitre
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 4 | 3 | 4
milligrams per decilitre | 0.72 (0.47) | 1.06 (0.36) | 1.03 (0.65)

11. Secondary Outcome: Serum Pyruvate
Time Frame: 24 hours post-operative
Population: Data were not collected for 5 participants in the Dexmedetomidine (Precedex®) arm. Data were not collected for 5 participants in the Propofol arm. Data were not collected for 3 participants in the Sevoflurane arm.
Measure: Mean (Standard Deviation); unit: milligrams per decilitre
Arm/Group | Dexmedetomidine (Precedex®) | Propofol | Sevoflurane
Number analyzed (Participants) | 2 | 1 | 3
milligrams per decilitre | 1.34 (0.85) | 1.32 (NA) — Standard Deviation not available since only 1 participant was analyzed for the assessment | 1.42 (0.69)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Sevoflurane | Dexmedetomidine (Precedex®) | Propofol
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 2/7 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sevoflurane (N=6) | Dexmedetomidine (Precedex®) (N=7) | Propofol (N=6)
Vomiting (General disorders) | 0 | 1 | 2
Fever (General disorders) | 2 | 1 | 0
lower back pain (General disorders) | 0 | 1 | 0
lethargy (General disorders) | 0 | 2 | 1
Nausea (General disorders) | 0 | 0 | 1
mood change (General disorders) | 1 | 1 | 0
feeding difficulties (General disorders) | 1 | 0 | 1
tachycardia (Cardiac disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT02053766/Prot_SAP_000.pdf